CLINICAL TRIAL: NCT04923867
Title: A Multicenter, Retrospective, Post-Market Clinical Follow-Up Study to Evaluate the Performance and Safety of Suturable DuraGen™
Brief Title: Suturable DuraGen™ PMCF Study
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C-DGSUT-001
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cerebrospinal Fluid Leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Supratentorial Procedure Group: Subjects that have undergone a supratentorial procedure with the use of Suturable DuraGen™.
  Interventions: Device: Suturable DuraGen™
- Infratentorial Procedure Group: Subjects that have undergone a infratentorial procedure with the use of Suturable DuraGen™.
  Interventions: Device: Suturable DuraGen™
- Spinal Procedure Group: Subjects that have undergone a spinal procedure with the use of Suturable DuraGen™.
  Interventions: Device: Suturable DuraGen™

INTERVENTIONS:
Device: Suturable DuraGen™ — Suturable DuraGen™ Dural Regeneration Matrix, an absorbable implant for repair of dural defects.

SUMMARY:
The primary goal of this study is to retrospectively collect data on the safety and efficacy of Suturable DuraGen™.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, non-interventional, retrospective Post-Market Clinical Follow-up (PMCF) study to evaluate the occurrence of post-operative cerebrospinal fluid (CSF) leaks within 30 days (and up to 90 days) after use of Suturable DuraGen™ for a supratentorial, infratentorial, or spinal procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 80 years of age
2. Subject has undergone either a supratentorial, an infratentorial, or a spinal procedure with the use of Suturable DuraGen™ prior to trial initiation
3. Availability of post-operative assessment results.

Exclusion Criteria:

1. There are no exclusionary criteria for this study population

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgery service in Hospital
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Patient Outcome | post-up to 90 days
  Occurrence of post-operative cerebrospinal fluid (CSF) leaks post-procedure

SECONDARY OUTCOMES:
Occurrence of Adverse Event | Between days 30-90
  Adverse event that occurred between days 30-90 post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tummon, Study Director — Integra LifeSciences
Locations (3):
- United States (3):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Baptist Medical Center, Jacksonville, Florida
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided